CLINICAL TRIAL: NCT06754007
Title: The Effectiveness of Rapid Optimisation of Performance Enhancement and Skill (ROPES) as an Exercise Training Programme for Sedentary Health Care Staff
Brief Title: Rapid Optimisation of Performance Enhancement and Skill (ROPES)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Singapore General Hospital (Other)
Responsible Party: Principal Investigator, Celia Tan Ia Choo, Senior Principal Physiotherapist, Singapore General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2024-3861
Record Dates: First submitted 2024-12-17; First posted 2024-12-31 (Actual); Last update posted 2025-02-14 (Actual); Status verified 2024-12

CONDITIONS: Sedentary Lifestyle
Keywords: Sedentary; healthcare workers
MeSH Terms: conditions — Sedentary Behavior

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control (No Intervention): 30 participants will be randomised into the CONTROL group and will continue to perform their normal activities. They will only be required to keep a log of their exercise intensity for each week over the 4-week period and record them on an online diary. The exercise log/diary consists of type of exercise, e.g. resistance or aerobic and duration of exercise session.
- ROPES (Experimental): The intervention is a 4-week training exercise program conducted by trained Physiotherapists.
  Interventions: Procedure: ROPES Training Programme

INTERVENTIONS:
Procedure: ROPES Training Programme — ROPES is a training programme that involves resistance training, whole-body exercises and HIIT aerobic sessions with each session lasting no longer than 45 minutes.
  Arms: ROPES

SUMMARY:
Despite innate knowledge of the benefits of regular physical activity, healthcare workers are just as physically inactive as the general population. Physical activity interventions delivered at the workplace seem perfect to improve the health of this large population.

The aim of the study is to deliver an efficacious, minimal time impost training program targeted at optimising health benefit while overcoming time-related barriers to initial uptake of regular exercise.

DETAILED DESCRIPTION:
To evaluate the effectiveness of a 4-week, easily accessible, time-optimised exercise program (ROPES - Rapid Optimisation of Performance Enhancement and Skill) for healthcare workers.

60 staff recruited from Singapore General Hospital (SGH) will be randomly assigned into 2 groups, CONTROL or ROPES group. The ratio to intervention and control group is at 1:1. The staff will be assigned to each group respectively.

ELIGIBILITY:
Inclusion Criteria:

* Age group: 21 - 70 years old
* All participants must be free of musculoskeletal, surgical and/or neurological injury in the past 6 months.
* Participants not engaged actively in regular exercise i.e. exercises less than once a week and at a duration less than 30 mins per session.
* Healthy with stable management of any existing diabetes, cholesterol and/or hypertension.
* They should have no issues with the Physical Activity Readiness Questionnaire (PAR-Q)

Exclusion Criteria:

* Participants under the age of 21 or over the age of 70
* Newly diagnosed diabetes/metabolic syndrome/high cholesterol or uncontrolled high BP >160 mmHg and under medical supervision.
* Subjects with cardiovascular conditions and on beta-blockers.
* Subjects who are pregnant or with recent (< 3 months) diagnosis of a medical condition, especially cardiac-related conditions.

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-01-02 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
Physical work capacity | From enrollment to the end of study at 8 weeks
  A standard physical work capacity test based on the linear relationship between heart rate, power output and oxygen consumption will estimate the work capacity.
  The higher the heart rate, the better the physical work capacity. Minimum value of heart rate is 155 bpm and maximum value is 199 bpm.

SECONDARY OUTCOMES:
Muscular Strength | From enrollment to the end of study at 8 weeks
  Handgrip strength will be measured using a hand-held dynamometer to determine functional strength.
BMI | From enrollment to the end of study at 8 weeks
  Height and weight will be measured on a body fat analyser and will be combined to report the BMI in kg/m^2.
Body Fat | From enrollment to the end of study at 8 weeks
  Body fat will be measured on a body composition analyser and will be reported in percentage %.

CONTACTS AND LOCATIONS:
Locations (1):
- Singapore General Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No